CLINICAL TRIAL: NCT05700825
Title: Rehabilitation of Airway Protection in Parkinson's Disease: Comparing In-person and Telehealth Service Delivery Models
Brief Title: Rehabilitation of Airway Protection in Parkinson's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Teachers College, Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Purdue University (Other)
Responsible Party: Principal Investigator, Michelle Troche, Professor, Principle Investigator, Teachers College, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NS126319; 1R01NS126319 (NIH)
Record Dates: First submitted 2022-12-22; First posted 2023-01-26 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease; Dysphagia
MeSH Terms: conditions — Parkinson Disease; Deglutition Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- In-person (Active Comparator)
  Interventions: Behavioral: Expiratory Muscle Strength Training + Cough Skill Training
- Telehealth (Experimental)
  Interventions: Behavioral: Expiratory Muscle Strength Training + Cough Skill Training

INTERVENTIONS:
Behavioral: Expiratory Muscle Strength Training + Cough Skill Training — Expiratory Muscle Strength Training (EMST). EMST is a widely used and efficacious treatment approach that uses a calibrated device with a one-way, spring-loaded pressure relief valve to mechanically overload the expiratory and submental muscles.
  Cough Skill Training (CST) involves a digital peak flow meter device which measures PEFR (peak expiratory flow rate) in liters/second and allows patients to receive immediate biofeedback.

SUMMARY:
Airway protective disorders are a prevalent and progressive consequence of Parkinson's Disease (PD), and often result in aspiration pneumonia which is the leading cause of death in PD. Despite this, a large number of patients with PD do not access specialized services to address these critical deficits. The investigators will examine the comparative effectiveness of a novel treatment paradigm delivered in-person versus via telehealth in persons with PD, as well as the role of patient burden and treatment adherence on outcomes; thus, the proposed research is relevant to public health and in line with NIH's mission to identify novel, efficacious, and accessible rehabilitation strategies for short- and long-term improvement of dysfunctional airway protection in PD.

DETAILED DESCRIPTION:
Progressive disorders of airway protection, such as swallowing disorders (dysphagia) and cough disorders (dystussia), are highly prevalent in PD and have significant negative implications for health and quality of life. In fact, aspiration pneumonia, commonly associated with dysphagia/dystussia, is a leading cause of death in PD. Despite this, there is currently no established standard of care for the treatment of airway protective disorders in this population. Even more critically, approximately 40% of individuals with PD in the United States do not access rehabilitation services or receive specialized care for these potentially life-threatening airway protective deficits. Expiratory Muscle Strength Training (EMST) and Cough Skill Training (CST) have been found to improve airway protective disorders in PD and be feasible via telehealth. However, a significant clinical-research gap remains in that it has not been demonstrated that clinical outcomes are comparable (non-inferior) when these treatments are delivered via telehealth versus in-person. This gap limits access to these important services with detrimental effects to health and quality of life. The long-term goal of this line of research is to improve the health outcomes of individuals with PD, specifically as they relate to airway protective dysfunction. The objective of this application is to pair EMST + CST - and compare clinical and patient-centered outcomes when conducted in-person versus via telehealth in the short- and the long-term. Also, the investigators will assess the role of specific patient burden factors and resultant treatment adherence on clinical outcomes. Therefore, the aims of this study are to: 1) Compare clinical and patient-centered outcomes following four weeks of intensive in-person vs. telehealth EMST+CST treatment in persons with PD, 2) Compare clinical and patient-centered outcomes from a long-term EMST+CST maintenance program offered in-person vs. via telehealth in persons with PD, and 3) Identify the role of specific patient burden factors (i.e., geographic location, cognitive function, disease severity, and caregiver burden) on treatment adherence in the short- and long-term and the influence of treatment adherence on clinical outcomes. The investigators will achieve these aims by conducting a two-arm, two site, randomized clinical trial in 120 people with PD comparing in-person vs. telehealth EMST+CST treatment after a four-week intensive period (aim1) and after a one year maintenance treatment period (with assessments at six and 12 months - aim 2). The investigators anticipate our findings will result in immediately translatable clinical deliverables that will have broad impact for reduced burden and improved accessibility of treatment. Further, these findings will inform our future studies investigating these treatments and service delivery models on long-term outcomes (i.e., aspiration pneumonia, hospitalization, death), accessibility, and healthcare costs.

ELIGIBILITY:
Inclusion criteria:

* Diagnosed with PD (Hoehn and Yahr Stages II-IV)126,127 confirmed by a Movement Disorders fellowship trained neurologist having reviewed the video recorded Movement Disorders Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) assessment for each participant and using strict UK brain bank criteria
* airway protective deficits as defined as a minimum of penetration of thin liquids (penetration-aspiration score>3) as determined by instrumental swallowing assessment and/or dystussia as determined by voluntary cough assessment (PEFR ≤4.1 L/s)
* not actively receiving exercise-based swallowing therapy
* between the ages of 50 and 90.

Exclusion criteria:

* Other neurological disorders (e.g., multiple sclerosis, stroke, brain tumor, etc.)
* history of head and neck cancer
* history of breathing disorders or diseases (e.g., COPD)
* history of smoking in the last five years
* uncontrolled hypertension
* difficulty complying due to neuropsychological dysfunction (i.e., severe depression with >28 on the Beck Depression Index (BDI-II), dementia with <19 on the Montreal Cognitive Assessment (MoCA))
* allergy to capsaicin or barium
* further than 1.5 hours (door to door) distance from either Teachers College, Columbia University or Purdue University.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Peak Expiratory Flow Rate (Cough PEFR) - phase 1 | Pretraining to posttraining (after four weeks of intensive training)
Change in Peak Expiratory Flow Rate (Cough PEFR) - phase 2 | post-training to post one-year maintenance
Change in Penetration-Aspiration Scale (PAS) - phase 1 | Pretraining to posttraining (after four weeks of intensive training)
  PAS, max value: 8 (most impaired), min value 1 (least impaired).
Change in Penetration-Aspiration Scale (PAS) - phase 2 | post-training to post one-year maintenance
  PAS, max value: 8 (most impaired), min value 1 (least impaired).

SECONDARY OUTCOMES:
Change in Maximum Expiratory Pressure - phase 1 | Pretraining to posttraining (after four weeks of intensive training)
Change in Maximum Expiratory Pressure - phase 2 | post-training to post one-year maintenance
Change in Cough expired volume - phase 1 | Pretraining to posttraining (after four weeks of intensive training)
Change in Cough expired volume - phase 2 | post-training to post one-year maintenance
Treatment Adherence - phase 1 | posttraining (after four weeks of intensive training)
  percent of prescribed training coughs and breaths completed
Change in Treatment Adherence- phase 2 | post-training to post one-year maintenance
  percent of prescribed training coughs and breaths completed
Change in SWAL-QOL- phase 1 | Pretraining to posttraining (after four weeks of intensive training)
  self-report questionnaire of swallowing quality of life, 44 min score, 220 max score - higher score is better QOL
Change in SWAL-QOL - phase 2 | post-training to post one-year maintenance
  self-report questionnaire of swallowing quality of life, 44 min score, 220 max score - higher score is better QOL

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Troche, PhD, Principal Investigator — Teachers College, Columbia University
Locations (2):
- United States (2):
  - Purdue University, West Lafayette, Indiana
  - Teachers College, Columbia University, New York, New York

IPD SHARING:
Plan to Share IPD: Yes